CLINICAL TRIAL: NCT04564755
Title: ABROCITINIB EXPANDED ACCESS PROTOCOL FOR THE TREATMENT OF ADOLESCENTS AND ADULTS WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: Abrocitinib Expanded Access Protocol in Adolescents and Adults With Moderate to Severe Atopic Dermatitis
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7451064; 2020-003610-12 (EudraCT Number); JADE REAL (Other: Alias Study Number)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema; expanded access
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — abrocitinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: abrocitinib — Participants will receive abrocitinib 100 mg or 200 mg orally once a day as directed by the investigator's clinical judgement

SUMMARY:
This is a multi-center, expanded access protocol to provide access to the investigational product, abrocitinib, to adolescent and adult patients with moderate to severe atopic dermatitis who have inadequate treatment options with available and approved medicated topical and systemic therapies and who are otherwise ineligible for participation in clinical studies with abrocitinib.

DETAILED DESCRIPTION:
This is a multi-center expanded access protocol (EAP) for the treatment of up to approximately 500 adult and adolescent (defined as age < 18 years) patients with moderate to severe atopic dermatitis for whom standard, approved medicated topical and systemic treatment options are inadequate and who would be suitable candidates for a trial of abrocitinib for potential treatment of moderate to severe atopic dermatitis. The study will also collect safety and exploratory efficacy data. Participants who meet the inclusion criteria and none of the exclusion criteria may be enrolled into the EAP to receive open-label oral treatment with abrocitinib.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* Clinical diagnosis of chronic atopic dermatitis for at least 6 months
* Inadequate treatment options with available, approved medicated topical and systemic therapies for moderate to severe atopic dermatitis
* Moderate to severe atopic dermatitis as indicated by at least one of the following: IGA ≥3; EASI ≥16
* Not eligible for participation in any ongoing clinical trial of abrocitinib, including lack of access due to geographical limitations

Exclusion Criteria:

* Medical, psychiatric, or laboratory abnormality that may increase the risk associated with study participation
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, malignancies, current or history of certain infections, lymphoproliferative disorders and other medical conditions at the discretion of the investigator
* Require treatment with prohibited medications during the study
* Discontinued prior treatment with any systemic JAK inhibitor due to safety or tolerability issues
* 12 to <18 years old without documented evidence of having received at least one dose of the varicella vaccine or without evidence of prior exposure to varicella zoster virus based on serological test
* Pregnant or breastfeeding women or women of childbearing potential who are sexually active and unwilling to use contraception

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (56):
- United States (21):
  - Cahaba Dermatology and Skin Health Center, Birmingham, Alabama
  - Antelope Valley Clinical Trials, Lancaster, California
  - Allergy & Asthma Care Center, Long Beach, California
  - Beach Allergy and Asthma Specialty Group, A Medical Corporation, Long Beach, California
  - ACRC Studies, San Diego, California
  - Palm Beach Dermatology, Delray Beach, Florida
  - Skin Care Research, Hollywood, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Dundee Dermatology, West Dundee, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - Bluegrass Allergy Research, Lexington, Kentucky
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - Bexley Dermatology Research, Bexley, Ohio
  - Hightower Clinical Trial Services - Lam Dermatology, Norman, Oklahoma
  - Health Concepts, Rapid City, South Dakota
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Memphis, Tennessee
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Houston Medical Imaging, Houston, Texas
  - West Virginia Research Institute, Morgantown, West Virginia
- Australia (6):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Dr Rodney Sinclair Pty Ltd, Melbourne, Victoria
  - Sinclair Dermatology, Melbourne, Victoria
  - Paratus Clinical Research Woden, Philip
- Austria (2):
  - Medizinische Universität Wien, Vienna, Vienna
  - Medical University of Vienna, Vienna
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Grand Hôpital de Charleroi, Loverval
- Canada (5):
  - Dermatology Research Institute, Calgary, Alberta
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Centre de recherche Saint-Louis, Québec
- Greece (3):
  - 401 General Military Hospital of Athens, Athens, Attikí
  - University General Hospital "ATTIKON", Athens, Attikí
  - "Ippokrateio" General Hospital of Thessaloniki interconnected with Hospital of Dermatology and Vener, Thessaloniki, Kentrikí Makedonía
- Centro de Dermatologia de Monterrey, Monterrey, Nuevo León, Mexico
- Universitair Medisch Centrum (UMCU) Utrecht, Utrecht, Netherlands
- NRC Institute of Immunology FMBA of Russia, Moscow, Russia
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, LAS Palmas
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario de Pontevedra Centro de Especialidades de Mollabao, Pontevedra
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Switzerland (5):
  - Universitätsspital Zürich, Zurich, Canton of Zurich
  - Inselspital, Universitätsklinik für Dermatologie, Bern
  - Inselspital, Universitätsspital Bern (Radiology), Bern
  - University Hospital Geneva, Geneva
  - Universitätsspital Zürich, Zurich
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451064